CLINICAL TRIAL: NCT05243329
Title: Investigating the Therapeutic Effects of Psilocybin in Treatment-Resistant Post-Traumatic Stress Disorder
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Halucenex Life Sciences Inc. (Industry)
Collaborators: KGK Science Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 22HLCPP01/HCX-2020-001
Record Dates: First submitted 2021-12-15; First posted 2022-02-17 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Treatment Resistant Disorders; Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Psilocybin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Psilocybin treatment for treatment-resistant PTSD (Experimental): Experimental Treatment:
  Experimental: Psilocybin
  10mg (low dose) on Day 7
  25mg (high dose) on Day 14
  10mg dose (optional top-up low dose) at Month 7
  Treatment Description:
  Drug: Psilocybin drug product suspension
  Psilocybin is manufactured as a bulk API powder. The psilocybin drug product suspension is prepared by a compounding pharmacist at the clinic site. The psilocybin drug product suspension will be mixed in a glass with water to produce the psilocybin solution for oral consumption. Subjects will be instructed to orally consume the study medication in the glass in its entirety.
  Psilocybin will be administered in the following doses and at the following time points for this study:
  * 1 mL of 10mg/mL (low dose) on Day 7 (10 mg)
  * 2.5 mL of 10 mg/mL (high dose) on Day 14 (25 mg)
  * [Optional dose] 1 mL of 10mg/mL (low dose) on Month 7/Day 210 (10 mg)
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — 10 mg or 25 mg oral aqueous psilocybin solution

SUMMARY:
Post-traumatic stress disorder (PTSD) is a complex disorder expressed as a variety of neurobiological symptoms, including anxiety, re-experiencing, hyperarousal, and avoidance symptoms, along with comorbidities such as anxiety, depression, and increased risk for self-medicating substance abuse. Currently, there are only two approved medications in the United States (US) for PTSD, paroxetine and sertraline.

Psychedelic medications, including psilocybin, have recently received breakthrough designation by the US Food and Drug Administration (FDA) for other psychiatric indications. Although no formal clinical trials have yet investigated psychedelic substances for the treatment of PTSD, the available evidence warrants such an investigation. The present study aims to investigate the effect of psilocybin on treatment-resistant PTSD.

DETAILED DESCRIPTION:
Post-traumatic stress disorder (PTSD) is a complex disorder expressed as a variety of neurobiological symptoms, including anxiety, re-experiencing, hyperarousal, and avoidance symptoms, along with comorbidities such as anxiety, depression, and increased risk for self-medicating substance abuse. Currently, there are only two approved medications in the United States (US) for PTSD, paroxetine and sertraline. These selective serotonin reuptake inhibitors (SSRIs) have limited efficacy. Furthermore, there is a lack of efficacious pharmacotherapy for treatment-resistant PTSD; PTSD remains a chronic and sometimes debilitating condition. New research into other treatment options for PTSD are warranted.

Psychedelic medications, including psilocybin, have recently received breakthrough designation by the US Food and Drug Administration (FDA) for other psychiatric indications. Psilocybin has received breakthrough designation for treatment of depression. Research on psilocybin has shown that it facilitates fear extinction in mice and promotes neuroplasticity, increasing neurogenesis, spinogenesis and synaptogenesis. These properties may contribute to antidepressive and anxiolytic effects. Psilocybin also reduces activity in the amygdala during threat responses; decreased amygdala reactivity is correlated with positive mood. This is particularly relevant since individuals with PTSD showed increased reactivity in the amygdala, which may increase the ability to process traumatic memories. Although no formal clinical trials have yet investigated psychedelic substances for the treatment of PTSD, the available evidence warrants such an investigation. The present study aims to investigate the effect of psilocybin on treatment-resistant PTSD.

ELIGIBILITY:
Inclusion Criteria:

- After signing and dating the informed consent documents, subject eligibility will be assessed. Subjects must meet the following criteria to be eligible for enrollment into the study.

1. Subjects must be ≥18 and ≤70 years of age.
2. Subjects must meet the Diagnostic & Statistical Manual of Mental Disorders - Version V (DSM-V) criteria for TR-PTSD.
3. Subjects must have treatment-resistant PTSD symptoms, defined as a CAPS score of ≥30 (signifying moderate to severe symptoms) following at least 3 months of prior SSRI or serotonin-norepinephrine reuptake inhibitor (SNRI) treatment in addition to at least 4 months of psychotherapy (adapted from Mithoefer et al, 2011).
4. Subjects must be able to communicate in English.

Exclusion Criteria:

* Subjects meeting any of the following criteria will not be eligible for participation in the study:

  1. Pregnant individuals and those of childbearing age not using effective contraception (e.g., oral contraceptive pill, injection, implant, patch, vaginal ring, intrauterine coil, intrauterine device, tubal ligation, or barrier method).
  2. Uncontrolled hypertension or BP ≥140/90 mmHg over 2 days, with at least 4 BP assessments completed.
  3. In the clinical judgement of the investigator, any hazard-posing medical, emotional, or significant character disorder or condition rendering unsuitability for the study. For example, poorly controlled diabetes, severe cardiovascular disease, seizure disorders, sleep apnea disorders (suspected or ineffectively treated), untrustworthiness, suicidality, etc.
  4. Any use of methamphetamines or any injection drug abuse in the past 30 days and/or a positive test for drugs of abuse (e.g., cocaine, amphetamines, opiates, benzodiazepines, etc.).
  5. Any other significant substance use disorder that may interfere with study objectives including consuming >5 cups of caffeinated coffee a day or inability, without discomfort, to refrain from smoking cigarettes or cannabis, or consuming alcohol for 7 hours.
  6. Blood draw or needle phobia.
  7. Suicidal attempt or active ideation deemed to present risk of suicide as judged by study clinical staff in past 30 days..
  8. BMI <14 or >42 or the Qualified investigator deems the patient sufficiently healthy to participate.
  9. Current or previously diagnosed schizophrenia spectrum or other psychotic disorders, including schizophrenia, schizoaffective disorder, schizotypal disorder, schizophreniform disorder or brief psychotic disorder; current or previous history of bipolar disorder, or obsessive-compulsive disorder.
  10. Any uncontrolled eating disorder (e.g., purging or anorexia or worsening of directionally undesirable weight change of 5 kg in past 30 days).
  11. Subjects with a diagnosis of DSM-5 personality disorder which has a major impact on the subject's current psychiatric status
  12. Use of any investigational drug, hallucinogen, or ketamine/esketamine within the past 30 days, or plan to use during the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-10-03 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Primary efficacy of psilocybin using the 11-Dimension Altered States of Consciousness (11D-ASC) will assess | Day 14
  This is a 42 item questionnaire assessing patient-rated subjective intensity of psilocybin's effects
PTSD symptom severity as measured by the Clinician-Administered PTSD Scale (CAPS-5) | Screening to 12 months follow up
  Total CAPS-5 Scores range from 0-80. Higher scores indicate greater symptom severity.
PTSD symptom severity as measured by the Posttraumatic Checklist for the DSM-5 (PCL-5) | Screening to 12 months follow up
  Total PCL-5 Scores range from 0-80. Higher scores indicate greater symptom severity.
Subjective distress caused by traumatic events as measured by the Impact of Events Scale Revised (IES-R). | Screening to 12 months follow up
  The IES-R is a 22-item self-report measure where respondents are asked to identify a specific stressful life event and then indicate how much they were distressed or bothered during the past seven days by each "difficulty" listed. Items are rated on a 5-point scale ranging from 0 ("not at all") to 4 ("extremely"). The IES-R yields a total score (ranging from 0 to 88).
Symptoms of Psychopathology as measured by the Symptom Checklist 90-R (SC90-R). | Screening to 12 months follow up
  The 90 items in the SC90-R are assessed by the subject using a 5-point rating scale.
Symptom severity, treatment response, and the efficacy of treatment studies of patients with mental disorders as measured by the Clinical Global Impression - Improvement (CGI-I)/ Clinical Global Impression - Severity (CGI-S). | Day 22
  The CGI-S scale is a 7-point, clinician-rated scale (ranging from 1 to 7, with 1 indicating a "normal state" and 7 indicating "among the most extremely ill patients").

SECONDARY OUTCOMES:
Anxiety as measured by the Beck Anxiety Inventory (BAI). | Up to 12 month follow up
  The BAI is a 21-item self-report inventor. Total BAI Scores range from 0-63; higher scores indicate more severe anxiety.
Anxiety as measured by the State Trait Anxiety Inventory - Trait Version (STAI-T). | Up to 6 month follow up
  The STAI-T scale consists of 20 items on a 4-point scale; Higher scores indicate greater anxiety.
Depression as measured by the Beck Depression Inventory (BDI). | Up to 12 month follow up
  The BDI is a 21-item, self-report rating inventory with each item scored on a scale value of 0 to 3; higher total scores indicating more severe depression symptoms.
Depression as measured by the Quick Inventory of Depressive Symptomatology - Self Report (QIDS-SR). | Up to 12 month follow up
  The QIDS-SR contains 16 items, with each item scored from 0 to 3.
Impairments in daily living as measured by the Sheehan Disability Scale (SDS). | Up to 12 month follow up
  This is a 3-item, clinician administered questionnaire with all items rated on an 11-point continuum, with higher scores indicating more severe impairment. (0 meaning "no impairment" to 10 meaning "most severe").
Body Mass Index (BMI) | Up to 12 month follow up
  Measure of body mass based on height and weight
Trauma Related Nightmare Survey | Up to 12 month follow up
  trauma-focused survey to track sleep and nightmare-related information

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Batten, PhD, Study Director — Halucenex Life Sciences; Paige Stevens, MD, Principal Investigator — Contracted
Locations (1):
- Halucenex Life Sciences Inc., Windsor, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No